CLINICAL TRIAL: NCT01968239
Title: A Randomized, Controlled Interventional Phase 2b (Proof of Concept) Study of the Efficacy, Safety, and Tolerability of Repeated Intravitreal Administration of Ranibizumab Guided by Morphological Changes Documented by Optical Coherence Tomography (OCT) in Subjects With Macular Edema Secondary to Branch Retinal Vein Occlusion (BRVO)
Brief Title: Proof of Concept Study of Re-treatment in BRVO With Ranibizumab Guided by OCT
Acronym: RabOCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, PD Dr. habil. Matus Rehak, MD, Ph.D, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201200543910
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: BRVO; Macular edema; Ranibizumab; re-treatment
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCT guided group (Experimental): Patients randomized to this group will get the intravitreal injection of 0.5 mg ranibizumab if the morphological macular changes for recurrence of macular edema (microcystic changes with or without increase of central retinal thickness) will be detected by OCT.
  Interventions: Drug: Ranibizumab
- Standard treatment (Active Comparator): Patients randomized to this group will get the intravitreal injection of 0.5 mg ranibizumab according to the in SmPC defined re-treatment criteria (re-injection if decrease of BCVA will be detected).
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — comparison of different re-treatment criteria for intravitreal injection of ranibizumab

SUMMARY:
The aim of the trial is to evaluate the efficacy and safety of intravitreal injections of ranibizumab for the treatment of macular edema due to BRVO if the re-treatment regimen is guided by morphological macular changes detected by OCT compared to re-treatment according to SmPC defined re-treatment criteria (in case of increase of CRT and concomitant decrease of BCVA).

DETAILED DESCRIPTION:
In a prospective, randomized, interventional, controlled phase IIb clinical the functional results of treatment with ranibizumab in patients with macular edema due to branch retinal vein occlusion when given according to morphological changes detected by OCT compared to standard re-treatment criteria according to SmPC

ELIGIBILITY:
Inclusion Criteria:

* Recurrence of macular edema defined as any kind of fluid accumulation in the macula (microcystic changes with or without increase of central retinal thickness) detected by OCT in the month 1 to 6 after the last Lucentis injection without any decrease of BCVA measured with ETDRS charts 2. Diagnosis of BRVO with macular edema treated with at least three intravitreally applied injections of ranibizumab after the up-load phase of treatment 3. Age ≥ 18 years 4. Ability and willingness to attend all scheduled visits and assessments 5. For sexually active women of childbearing potential, use of an appropriate form of contraception (or abstinence) for the duration of the study

Exclusion Criteria:

1. Macular edema due to another etiology than retinal vein occlusion (e.g. diabetic maculopathy, uveitis, age related macular degeneration, Irvine-Gass syndrome)
2. Evidence upon examination of vitreoretinal interface disease (e.g., vitreomacular traction, epiretinal membrane), either on clinical examination or OCT, thought to be contributing to macular edema
3. Use of intraocular or periocular injection of steroids in the study eye (e.g., triamcinolone) prior to study entry
4. History of cerebral vascular accident, myocardial infarction, transient ischemic attacks in last 6 months
5. Pregnancy (positive pregnancy test) or lactation
6. History of allergy to humanized antibodies or any component of the ranibizumab formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-06-17 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
change of best corrected visual acuity (BCVA) measured in ETDRS letters | 12 months

SECONDARY OUTCOMES:
Central retinal thickness (CRT) | 12 months
Number of applied ranibizumab injections | 12 months
• Rates of patients developing a neovascularisation of the retina/ anterior segment | 12 months
Assessment of safety: serious adverse events/ reactions; AEs/ARs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matus Rehak, MD, Ph.D., Principal Investigator — Department of Ophthalmology, University of Leipzig, Germany
Locations (1):
- Department of Ophthalmology, University Leipzig, Leipzig, Germany